CLINICAL TRIAL: NCT07146412
Title: Impact of a Multimodal Lifestyle Intervention on Dementia Risk Factors and Attitude Related to Dementia Risk: A Logistical Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HudsonAlpha Institute for Biotechnology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 0124
Record Dates: First submitted 2025-08-15; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Cognitive Impairment; Alzheimer Blood Biomarkers; Alzheimer Disease (AD); Mild Cognitive Impairment (MCI)
Keywords: alzheimer; cognitive impairment; APOE; PRS; pTau217
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Not high risk for conversion to cognitive impairment (No Intervention): This group will be defined by individuals who are not high risk by our study-defined rubric taking family history, Apolipoprotein E (APOE) genotype, Alzheimer's disease (AD) polygenic risk score (PRS), modified Cardiovascular Risk Factors, Aging and Incidence of Dementia (mCAIDE) score, lifestyle score described by Dhana and colleauges (see references section), Montreal Cognitive Assessment (MoCA), self-reported race/ethnicity, and pTau217 level into account.
- High risk for conversion to cognitive impairment (Experimental): This group will be defined by individuals who are high risk by our study-defined rubric taking family history, APOE genotype, AD PRS, mCAIDE score, lifestyle score described by Dhana and colleauges (see references section), MoCA, self-reported race/ethnicity, and pTau217 level into account. Individuals in this group will be offered a multimodal lifestyle intervention targeting the prevention of cognitive decline based on previous studies of lifestyle interventions for the prevention or delay of dementia as described in previous studies (see references section).
  Interventions: Behavioral: Multimodal Lifestyle Intervention

INTERVENTIONS:
Behavioral: Multimodal Lifestyle Intervention — The intervention supports adoption and maintenance of healthy behaviors including healthy nutrition The Mediterranean-DASH (Dietary Approaches to Stop Hypertension) Intervention for Neurodegenerative Delay, or MIND Diet), physical activity (150 min/week of moderate activity), stress management, weight management, and adherence to doctor-prescribed medical regimens. In addition, participants will be encouraged to participate regularly in social and learning activities, and to engage in cognitive training via Posit's BrainHQ web-based training tools (brainhq.com). Participants will be supported by telephone-based health coaching. Coaches will be currently licensed allied health providers such as Registered Dietitians. Using the combination of an individual's biological data (including genomics, blood, stool, saliva, etc.), activity data, behavioral data, and other incoming streams of health information, the coach will tailor the lifestyle intervention for each participant.
  Arms: High risk for conversion to cognitive impairment

SUMMARY:
Many individuals develop dementia, and dementia has multiple causes, yet we currently have limited treatment options. A critical observation of the effectiveness of the available dementia treatments is that they tend to be more effective when started early. Previous studies have shown that multimodal lifestyle interventions can significantly delay the onset of Alzheimer's dementia in individuals with high risk for Alzheimer's or with Mild Cognitive Impairment (MCI). These interventions may be less effective when initiated after dementia has already been diagnosed or is more advanced.

This study has two primary goals. The first goal is to assess attitudes around dementia risk for participants throughout the study as they learn of their personalized risk and possible lifestyle factors that may modify that risk. The second goal is to serve as a logistical pilot for the implementation of data collection and processing and multimodal lifestyle intervention to reduce the risk factors of dementia in individuals without current cognitive impairment but who are at high risk of progression to dementia. Secondary goals of this study include better defining what factors contribute the most risk to dementia and identifying sub-types of dementia defined by different genetic and molecular risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Adults 65-75 years of age at enrollment with at least one self-reported 1st-degree relative who had or has any kind of dementia
* Montreal Cognitive Assessment (MoCA) score > 24 at initial enrollment
* Able and willing to comprehend and sign the informed consent document
* Able and willing to perform required physical performance tests
* Able and willing to provide the study's minimum samples
* Able and willing to conduct the study's minimum procedures
* Able and willing to complete surveys, cognitive assessments, and questionnaires in English only
* Has or has ready access to a PC, tablet, or smartphone with an internet connection required for procedures that they consent to

Exclusion Criteria:

* A diagnosis of cognitive impairment of any kind, including Alzheimer's disease, mild cognitive impairment, or any other diagnosis of dementia
* If a subject is found to have cognitive impairment at initial enrollment (Montreal Cognitive Assessment (MoCA) score<25), they will be excluded from the study
* Self-reported pregnancy
* Children under 19 years of age
* Individuals not fluent in written and spoken English
* Self-reported chronic or end-stage disease that would interfere with their participation in the study
* Hospitalization for any reason in the past 3 months
* Severe hearing and visual impairment that would interfere with the ability to complete study measures
* Any other vulnerable subject at the time of enrollment as specified above

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-05-02 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Attitudes around dementia risk for participants throughout the study as they learn of their personalized risk and possible lifestyle factors that may modify that risk. | At enrollment (week -26 to week -4), at return of results visit indicating level of dementia risk (week 0), and (for participant that qualify for the multimodal lifestyle intervention arm) at week 26.
  All participants will be offered a survey about perception of and attitudes toward dementia risk using the scaling strategy described by Kasparian and colleagues and dementia questions from Kim and colleagues (see references).
REVEAL Impact of Genetics Testing in Alzheimer's Disease Distress Subscale | Week 1 and Week 26 (1 week after return of results visit, and also at final site visit).
  Participants identified as high risk (multimodal lifestyle intervention arm) will be asked to complete the REVEAL (Risk Evaluation and Education for Alzheimer's Disease) Impact of Genetics Testing in Alzheimer's Disease (IGT-AD) Distress Subscale. The scale is 12 items on a Likert scale, with higher scores indicating more distress.

SECONDARY OUTCOMES:
pTau217 level | Measured at screening (week -26 to -4), and, for high risk participants, at enrollment for intervention (week 0) as well as at 26 weeks into completing a multimodal lifestyle intervention.
  Level of pTau217 (picograms/milliliter, pg/mL). Limit of quantification 0.06 pg/mL, assay detection limit 0.03 pg/mL, threshold >0.18 pg/mL indicated as a surrogate marker for beta amyloid pathology, no upper bound specified by testing lab (labcorp). Higher scores indicate a worse outcome.
MoCA score | Measured at screening (week -26 to -4), and, for high risk participants, at enrollment for intervention (week 0) as well as at 26 weeks into completing a multimodal lifestyle intervention.
  Montreal Cognitive Assessment. Range 0-30. Lower scores correlate with more cognitive impairment. Study threshold for possible mild cognitive impairment (MCI) set at <25, but in this secondary outcome measure MoCA score will be evaluated as a continuous value. Lower scores indicate a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Smith Family Clinic for Genomic Medicine, Huntsville, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
All available IPD will be shared with qualified researchers under controlled access.
Supporting Information: Study Protocol, ICF
Time Frame: IPD and supporting information will be available upon initial publication describing the final study results.
Access Criteria: IPD will be made available to qualified researchers under controlled access. They will be able to access all available de-identified data.

REFERENCES:
- [Background] Chung WW, Chen CA, Cupples LA, Roberts JS, Hiraki SC, Nair AK, Green RC, Stern RA. A new scale measuring psychologic impact of genetic susceptibility testing for Alzheimer disease. Alzheimer Dis Assoc Disord. 2009 Jan-Mar;23(1):50-6. doi: 10.1097/wad.0b013e318188429e. PMID 19266699
- [Background] Kim S, Sargent-Cox K, Cherbuin N, Anstey KJ. Development of the motivation to change lifestyle and health behaviours for dementia risk reduction scale. Dement Geriatr Cogn Dis Extra. 2014 Jun 5;4(2):172-83. doi: 10.1159/000362228. eCollection 2014 May. PMID 25028583
- [Background] Kasparian NA, Wakefield CE, Meiser B. Assessment of psychosocial outcomes in genetic counseling research: an overview of available measurement scales. J Genet Couns. 2007 Dec;16(6):693-712. doi: 10.1007/s10897-007-9111-6. Epub 2007 Aug 13. PMID 17694397
- [Background] Baker LD, Espeland MA, Whitmer RA, Snyder HM, Leng X, Lovato L, Papp KV, Yu M, Kivipelto M, Alexander AS, Antkowiak S, Cleveland M, Day C, Elbein R, Tomaszewski Farias S, Felton D, Garcia KR, Gitelman DR, Graef S, Howard M, Katula J, Lambert K, Matongo O, McDonald AM, Pavlik V, Raman R, Salloway S, Tangney C, Ventrelle J, Wilmoth S, Willliams BJ, Wing R, Woolard N, Carrillo MC. Structured vs Self-Guided Multidomain Lifestyle Interventions for Global Cognitive Function: The US POINTER Randomized Clinical Trial. JAMA. 2025 Aug 26;334(8):681-691. doi: 10.1001/jama.2025.12923. PMID 40720610
- [Background] Ornish D, Madison C, Kivipelto M, Kemp C, McCulloch CE, Galasko D, Artz J, Rentz D, Lin J, Norman K, Ornish A, Tranter S, DeLamarter N, Wingers N, Richling C, Kaddurah-Daouk R, Knight R, McDonald D, Patel L, Verdin E, E Tanzi R, Arnold SE. Effects of intensive lifestyle changes on the progression of mild cognitive impairment or early dementia due to Alzheimer's disease: a randomized, controlled clinical trial. Alzheimers Res Ther. 2024 Jun 7;16(1):122. doi: 10.1186/s13195-024-01482-z. PMID 38849944
- [Background] Roach JC, Rapozo MK, Hara J, Glusman G, Lovejoy J, Shankle WR, Hood L; COCOA Consortium:. A Remotely Coached Multimodal Lifestyle Intervention for Alzheimer's Disease Ameliorates Functional and Cognitive Outcomes. J Alzheimers Dis. 2023;96(2):591-607. doi: 10.3233/JAD-230403. PMID 37840487
- [Background] Roach JC, Hara J, Fridman D, Lovejoy JC, Jade K, Heim L, Romansik R, Swietlikowski A, Phillips S, Rapozo MK, Shay MA, Fischer D, Funk C, Dill L, Brant-Zawadzki M, Hood L, Shankle WR. The Coaching for Cognition in Alzheimer's (COCOA) trial: Study design. Alzheimers Dement (N Y). 2022 Jul 26;8(1):e12318. doi: 10.1002/trc2.12318. eCollection 2022. PMID 35910672
- [Background] Kivipelto M, Solomon A, Ahtiluoto S, Ngandu T, Lehtisalo J, Antikainen R, Backman L, Hanninen T, Jula A, Laatikainen T, Lindstrom J, Mangialasche F, Nissinen A, Paajanen T, Pajala S, Peltonen M, Rauramaa R, Stigsdotter-Neely A, Strandberg T, Tuomilehto J, Soininen H. The Finnish Geriatric Intervention Study to Prevent Cognitive Impairment and Disability (FINGER): study design and progress. Alzheimers Dement. 2013 Nov;9(6):657-65. doi: 10.1016/j.jalz.2012.09.012. Epub 2013 Jan 17. PMID 23332672
- [Background] Dhana K, Evans DA, Rajan KB, Bennett DA, Morris MC. Healthy lifestyle and the risk of Alzheimer dementia: Findings from 2 longitudinal studies. Neurology. 2020 Jul 28;95(4):e374-e383. doi: 10.1212/WNL.0000000000009816. Epub 2020 Jun 17. PMID 32554763
- See also: Healthy Outcomes through Phenomic Exploration for Alzheimer's Disease — https://www.hudsonalpha.org/hopead/